CLINICAL TRIAL: NCT00039546
Title: 'tAnGo', A Phase III Randomised Trial Of Gemcitabine In Paclitaxel-Containing, Epirubicin-Based, Adjuvant Chemotherapy For ER/PgR-Poor, Early Stage, Breast Cancer
Brief Title: Combination Chemotherapy in Treating Women With Breast Cancer Who Have Undergone Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Research Campaign Clinical Trials Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CRC-TU-TANGO; CDR0000069396 (Registry Identifier: PDQ (Physician Data Query)); EU-20058
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2005-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Epirubicin; Gemcitabine; Paclitaxel; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: gemcitabine hydrochloride
Drug: paclitaxel
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which chemotherapy regimen is more effective in treating women after surgery for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of paclitaxel, epirubicin, and cyclophosphamide with or without gemcitabine in treating women who have undergone surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the 5-year and 10-year disease-free survival and overall survival of women with completely resected early stage breast cancer treated with adjuvant paclitaxel, epirubicin, and cyclophosphamide with or without gemcitabine.
* Compare the toxicity, dose-intensity, and tolerability of these regimens in these patients.
* Compare the serious adverse events in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to nodal status (negative vs 1-3 vs 4 or more), age (50 and under vs over 50), estrogen receptor status (negative vs weakly positive vs positive), concurrent radiotherapy (no vs yes), HER2 status (3+ overexpression vs other vs not measured), and country. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive epirubicin IV, cyclophosphamide IV, and paclitaxel IV over 3 hours on day 1. Patients also receive gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive epirubicin, cyclophosphamide, and paclitaxel as in arm I.

Patients are followed every 3 months for 6 months, every 6 months for 3 years, and then annually for 6 years.

PROJECTED ACCRUAL: A total of 3,000 patients (1,500 per treatment arm) will be accrued for this study within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed invasive breast cancer

  * Early stage disease
  * Completely resected disease

    * No more than 8 weeks since prior resection
* Any nodal status
* Indication for adjuvant chemotherapy
* No metastatic disease
* Hormone receptor status:

  * Estrogen receptor negative or weakly positive OR
  * Estrogen receptor positive AND progesterone receptor negative or weakly positive

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm3
* Platelet count greater than 100,000/mm3
* Hemoglobin greater than 9 g/dL

Hepatic:

* Bilirubin normal
* AST and ALT no greater than 1.5 times normal

Renal:

* Creatinine no greater than 1.5 times normal

Other:

* Fit to receive study chemotherapy
* No active uncontrolled infection
* No other malignancy within the past 10 years except basal cell carcinoma or carcinoma in situ of the cervix
* No other concurrent medical or psychiatric problems that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08

CONTACTS AND LOCATIONS:
Overall Officials: Helen Howard, PhD, Study Chair — Cancer Research Campaign Clinical Trials Centre
Locations (46):
- United Kingdom (46):
  - Queen Elizabeth Hospital at University of Birmingham, Birmingham, England
  - Cancer Research UK Clinical Trials Unit - Birmingham, Birmingham, England
  - City Hospital - Birmingham, Birmingham, England
  - Birmingham Heartlands and Solihull NHS Trust -Teaching, Birmingham, England
  - Queen's Hospital, Burton, Burton-on-Trent, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Broomfield Hospital, Chelmsford, Essex, England
  - Essex County Hospital, Colchester, England
  - Walsgrave Hospital, Coventry, England
  - Dorset County Hospital, Dorchester, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Princess Royal Hospital, Hull, England
  - Hinchingbrooke Hospital, Huntingdon, England
  - King George Hospital, Ilford, Essex, England
  - Crosshouse Hospital, Kilmarnock, England
  - Cookridge Hospital at Leeds Teaching Hospital NHS Trust, Leeds, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - St. George's Hospital, London, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Northampton General Hospital NHS Trust, Northampton, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Derriford Hospital, Plymouth, England
  - Oldchurch Hospital, Romford, England
  - Thornbury Hospital, Sheffield, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - West Suffolk Hospital, Suffolk, England
  - Torbay Hospital, Torquay Devon, England
  - Walsall Manor Hospital, Walsall, England
  - Sandwell General Hospital, West Bromwich, England
  - Good Hope Hospital Trust, West Midlands, England
  - Worcester Royal Hospital, Worcester, England
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland
  - Velindre Cancer Center at Velinde Hospital, Cardiff, Wales
  - Hairmyres Hospital, East Kilbride
  - Hull Royal Infirmary, Hull
  - Queen Elizabeth Hospital, Kings Lynn
  - Glan Clywd District General Hospital, Rhyl, Denbighshire
  - Singleton Hospital, Swansea
  - Morriston Hospital NHS Trust, West Glamorgen

REFERENCES:
- [Derived] Earl HM, Hiller L, Howard HC, Dunn JA, Young J, Bowden SJ, McDermaid M, Waterhouse AK, Wilson G, Agrawal R, O'Reilly S, Bowman A, Ritchie DM, Goodman A, Hickish T, McAdam K, Cameron D, Dodwell D, Rea DW, Caldas C, Provenzano E, Abraham JE, Canney P, Crown JP, Kennedy MJ, Coleman R, Leonard RC, Carmichael JA, Wardley AM, Poole CJ; tAnGo trial collaborators. Addition of gemcitabine to paclitaxel, epirubicin, and cyclophosphamide adjuvant chemotherapy for women with early-stage breast cancer (tAnGo): final 10-year follow-up of an open-label, randomised, phase 3 trial. Lancet Oncol. 2017 Jun;18(6):755-769. doi: 10.1016/S1470-2045(17)30319-4. Epub 2017 May 4. PMID 28479233